CLINICAL TRIAL: NCT02709473
Title: Does the Choice of Administration Sequence of Propofol and Remifentanil Affect the ED50 and ED95 of Rocuronium for Rapid Sequence Induction of Anesthesia?
Brief Title: The Effect of Propofol and Remifentanil Sequence on ED50 and ED95 of Rocuronium in Rapid Sequence Induction Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Menekse Ozcelik, MD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 31-31412
Record Dates: First submitted 2016-02-23; First posted 2016-03-16 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Anesthesia; Neuromuscular Blockade
Keywords: propofol; remifentanil; rocuronium
MeSH Terms: interventions — Propofol; Remifentanil; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Active Comparator): Propofol arm includes patients that induction of general anesthesia started with propofol and followed by remifentanil and rocuronium administration
  Interventions: Drug: Propofol; Drug: Remifentanil; Drug: Rocuronium
- remifentanil (Active Comparator): Remifentanil arm include patients that induction of general anesthesia started with remifentanil and followed by propofol and rocuronium administration
  Interventions: Drug: Propofol; Drug: Remifentanil; Drug: Rocuronium

INTERVENTIONS:
Drug: Propofol — Propofol will be used in either two arms. The injection sequence will be changed. In propofol arm of the study, general anesthesia will be started with 2 mg/kg propofol administered within 15 seconds. And, then remifentanil will be given. In remifentanil arm of the study, 2 mg/kg propofol will be applied within 15 seconds following remifentanil injection.
Drug: Remifentanil — Remifentanil will be used in either two arms. The injection sequence will be changed. In remifentanil arm, general anesthesia will be started with 2 μg/kg remifentanil administered within 30 seconds. And then propofol will be given. In propofol arm of the study the same dose will be applied within 30 seconds following propofol administration.
  Other Names: Ultiva
Drug: Rocuronium — Rocuronium will be used for either two study arms. Rocuronium will be given in a 0.8 mg/kg dosage in the first study subject. And then, if the intubation condition is acceptable, the dose of the rocuronium will be decreased by 0.1 mg/kg for the next patient. Otherwise, if the intubation condition is not acceptable, the rocuronium dosage will be increased by 0.1 mg/kg for the next patient. This will be continue for ten crossover points (the point that turn from unsuccessful intubation to successful intubation).
  Other Names: Esmeron

SUMMARY:
Rapid sequence induction (RSI) is a well-known procedure to maintain a safe and rapid airway in patients especially at risk of aspiration. Propofol and rocuronium are generally used agents for RSI. However, the difficult airway scenarios are always valid for these patients, even without predictive signs of difficult airway. Therefore, it is important to decrease the rocuronium dose used in RSI to achieve a rapid recovery of a neuromuscular conduction with the aid of a reversal agent in case of difficult airway. The short acting opioids such as remifentanil may be helpful to reduce the dose of rocuronium in RSI.

DETAILED DESCRIPTION:
Rapid sequence induction is a widely used anesthesia technique to achieve a safe airway control. However, the difficult airway may be expected in these patients as in the others. In the difficult airway situation, cholinesterase inhibitors and sugammadex may be used for the reversal. However, sugammadex is not always available due to its cost in every hospital. In addition to this, it is well-known that cholinesterase inhibitors do not work well in case of deep neuromuscular block. In consideration of these informations, the recovery of the neuromuscular block gain an importance in patients undergoing RSI with difficult airway. Therefore, decreasing the dosage of non-depolarizing neuromuscular agent may be helpful in case of the difficult airway situations. With the aim of decreasing the neuromuscular blocker dosage, opioid analgesics especially remifentanil is preferred combined with propofol to decrease the hemodynamic response to laryngoscopy and intubation. A recent study demonstrated that after induction of anesthesia with remifentanil and propofol, ED50 of rocuronium for acceptable intubation conditions was 0.20 mg/kg. In another study, the authors showed that the administration sequence of propofol and remifentanil for target controlled anesthesia affect the onset time of rocuronium due to change in cardiac output. The authors concluded that the prior administration of remifentanil decreased the cardiac output and delayed the onset time of rocuronium.

The investigators hypothesized that prior administration of remifentanil compared to propofol may increase the ED50 and ED95 of rocuronium for acceptable intubation conditions in RSI.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II patients
* patients scheduled for elective surgery

Exclusion Criteria:

* suspected or known difficult airway
* a significant renal or hepatic dysfunction
* a known neuromuscular disease
* hypertension
* a known allergy to one of the drugs used in general anesthesia
* a body mass index lower than 18.5 kg/m2 or higher than 30 kg/m2
* intake of any medication that might interact with rocuronium
* patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
ED50 of rocuronium | One minute after rocuronium injection
  ED50 of rocuronium means the dose of rocuronium that is required for providing acceptable intubation conditions in the 50% of patients undergoing intubation. Each individual dose that allow or not allow an acceptable intubation condition will determine the next patient rocuronium dose. At the end, ED50 of rocuronium will be calculated as means of drug dosage that providing acceptable intubation condition.
ED95 of rocuronium | One minute after rocuronium injection
  ED595 of rocuronium means the dose of rocuronium that is required for providing acceptable intubation conditions in the 95% of patients undergoing intubation. Each individual dose that allow or not allow an acceptable intubation condition will determine the next patient rocuronium dose. At the end, ED95 of rocuronium will be estimated by using statistical tools such as pava estimator or R code.

SECONDARY OUTCOMES:
mean arterial blood pressure | before and after 10 minutes of induction of anesthesia
  the effect of propofol and remifentanil administration sequence on mean arterial blood pressure will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Can, Assoc Prof, Study Director — Ankara University Department of Anesthesiology and Intensive Care Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University, Ankara
  - Harran University, Sanliurfa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh AY, Cho SJ, Seo KS, Ryu JH, Han SH, Hwang JW. Dose of rocuronium for rapid tracheal intubation following remifentanil 2 mug kg-1 and propofol 2 mg kg-1. Eur J Anaesthesiol. 2013 Sep;30(9):550-5. doi: 10.1097/EJA.0b013e3283622ba0. PMID 23698704
- [Background] Na HS, Hwang JW, Park SH, Oh AY, Park HP, Jeon YT, Do SH. Drug-administration sequence of target-controlled propofol and remifentanil influences the onset of rocuronium. A double-blind, randomized trial. Acta Anaesthesiol Scand. 2012 May;56(5):558-64. doi: 10.1111/j.1399-6576.2012.02648.x. Epub 2012 Feb 7. PMID 22313514
- [Background] Dewhirst E, Tobias JD, Martin DP. Propofol and remifentanil for rapid sequence intubation in a pediatric patient at risk for aspiration with elevated intracranial pressure. Pediatr Emerg Care. 2013 Nov;29(11):1201-3. doi: 10.1097/PEC.0b013e3182aa136d. PMID 24196089